CLINICAL TRIAL: NCT04989881
Title: Comparison of Dry-lab Laparoscopic Training and Robotic Virtual Simulator Training to Develop Basic Laparoscopic Skills: A Randomized Clinical Trial
Brief Title: Comparison of Dry-lab Laparoscopic Training and Robotic Virtual Simulator
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Pouya Iranmanesh, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: University of Geneva
Record Dates: First submitted 2021-04-07; First posted 2021-08-04 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Da Vinci Simulator (Experimental): Participants will undergo a single session of training using the da Vinci Simulator
  Interventions: Device: da Vinci Simulator
- Laparascopic training box (Active Comparator): Participants will undergo a single session of training using a laparoscopic training box
  Interventions: Device: Laparascopic training box

INTERVENTIONS:
Device: da Vinci Simulator — Single training session
  Arms: Da Vinci Simulator
Device: Laparascopic training box — Single training session
  Arms: Laparascopic training box

SUMMARY:
The objective of the present study is to compare the effectiveness of dry-lab laparoscopic training and robotic simulator training among medical students without any prior laparoscopic experience.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial conducted at the Swiss Foundation For Innovation And Training In Surgery (SFITS), which is part of the Geneva University Hospital in Switzerland. Recruitment of a sample of 100 medical students with no prior experience in laparoscopic surgery will be performed. The participants will be randomized in 2 groups (50 participants in each group). The study group will undergo a single session of training using a standard, dry-lab laparoscopic box. The control group will undergo a single session of training using the da Vinci Skills Simulator. Post-training surgical skills for both groups will be measured using exercises from the FLS manual skills assessment. The overall performance on the FLS test will be compared between the two groups .

ELIGIBILITY:
Inclusion Criteria:

* Medical student at the University of Geneva

Exclusion Criteria:

* Previous laparoscopic experience
* Stereoblindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
FLS score post-training session | Up to 1 hour after the beginning of the exam session.
  This score is a composite outcome combining the time needed to finish the exercises and the proficiency in performing them (number of dropped objects, lack of movements precision, exercises rules violations, etc.). The score will go from 0 (worst score) to 800 (best score), with a passing score of 356.

SECONDARY OUTCOMES:
Times needed to perform training exercises | Up to 1 hour after the beginning of the training session
  Time required to perform the training exercises will be measured in both groups (dry-lab laparoscopic box and da Vinci skills simulator)

CONTACTS AND LOCATIONS:
Overall Officials: Pouya Iranmanesh, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No